CLINICAL TRIAL: NCT07095335
Title: Evaluating the Effectiveness of Simulation Experiences to Help Navigate Racism and Hidden Bias
Brief Title: Evaluating Simulation Experiences to Help Navigate Racism and Hidden Bias
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Monakshi Sawhney, Associate Professor, Queen's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 6041616
Record Dates: First submitted 2025-05-18; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-06

CONDITIONS: Implicit Bias
Keywords: Implicit bias; racism; nurisng; clinical settings; nursing students; simulation experiences; education intervention
MeSH Terms: conditions — Bias, Implicit; Racism

STUDY DESIGN:
Intervention Model Description: Quasi-experimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): A-CHARM education and virtual simulation
  Interventions: Other: education intervention A-CHARM

INTERVENTIONS:
Other: education intervention A-CHARM — Didactic education plus virtual simulation regarding discrimination in the hospital setting

SUMMARY:
This study utilizes a quasi-experimental design to examine the acceptability, usability and impact of the A-CHARM resources including the pre-learning, the SEs and the debrief. Consenting participants will be asked to complete a demographic questionnaire and pre-simulation assessment of cultural humility using the Cultural Humility Scale, and cultural awareness using the Cultural Diversity Awareness Questionnaire. Participants will complete an education intervention that provides definitions of race, racism, and discrimination and provides an overview of the Six-Step Approach, ERASE framework and Microaggression Triangle model. Following the education intervention, they will complete a SE and a post-simulation questionnaire that reassess cultural humility, cultural awareness and the usability and acceptability of the SE.

DETAILED DESCRIPTION:
Background and Literature Review:

Anti-Black and anti-Asian racism has increased significantly since the COVID-19 pandemic, with the number of hate crimes committed due to race or ethnicity increasing by 80% in Canada in 2020. This includes police-reported hate crimes targeting the Black, East or Southeast Asian, Indigenous, and South Asian peoples. Healthcare providers, including nurses who are persons of color, are not exempt from experiencing racism and hidden biases. These experiences often occur in the clinical setting, are unreported or underreported, and have a negative impact on nurses. A study conducted with nurses (n= 788) in New Jersey, United States, examined the direct, indirect, and interactive effects of individual (race), interpersonal (workplace racial microaggressions), and institutional (racial climate) factors on hospital-based nurses' emotional well- being. Compared to White nurses, non-white nurses reported higher emotional distress, more negative racial climates, and more microaggressions due to race.

Nursing students who experience racism or inappropriate comments in the clinical setting often do not possess appropriate strategies regarding how to respond. In addition, faculty, colleagues or other bystanders may not know how to respond. Traditionally, the method of coping has been avoidance or silence.

However, by not addressing racism it can indicate that inappropriate behaviours are acceptable. Providing nursing students with opportunities to critically examine how they may navigate inappropriate comments or racism, if they experience or witness it, is one strategy that can be utilized. Simulation education provides an opportunity for nursing students to engage in scenarios that based on real life experiences in a safe environment. In this proposed study we utilize the term simulation experiences (SEs) to highlight the lived experiences that the simulations are based on.

Due to the lack of available resources an education session and five virtual simulation experiences (SEs) were developed through the A-CHARM (Addressing Culturally based Hidden bias and RacisM) nursing project.

A search of the literature for frameworks or steps that healthcare professionals, including nursing students, can use to address inappropriate comments or racism in the clinical setting was also conducted. Three models were found and include the: 1) Six-Step Approach, 2) ERASE framework 3) Microaggression Triangle model.

Nursing students and clinical faculty require the opportunity to practice using these frameworks in a safe environment prior to utilizing them in real world situations. Simulation experiences can be used to create a safe environment for nursing students to critically assess how they could us these frameworks to address hidden-bias and racism prior to experiencing or witnessing them. These SEs can be a great resource; however, they need to be evaluated.

Research question and objectives: The research question for this study is: In nursing students and clinical nursing faculty/instructors, what is the effectiveness of an education session and virtual simulation experiences (SE's) on cultural awareness and the ability to utilize strategies to navigate racism and inappropriate comments in the clinical setting.

The specific objectives are:

1. To describe the acceptability, and usability of the virtual simulation experiences (SEs) that focus on how to professionally address racism and inappropriate comments.
2. To examine the effect of the education intervention and the SEs on cultural humility and cultural awareness.

Method:

This cohort study utilizes a quasi-experimental design (quantitative and qualitative) to examine the acceptability, usability and impact of the A-CHARM resources including the pre-learning, the SEs and the debrief. Consenting participants will be asked to complete a demographic questionnaire and pre-simulation assessment of cultural humility using the Cultural Humility Scale, and cultural awareness using the Cultural Diversity Awareness Questionnaire.

Intervention: Participants will complete an education session that provides definitions of race, racism, and discrimination and provides an overview of the Six-Step Approach, ERASE framework and Microaggression Triangle model. Following the education session, they will complete a SE and a post-simulation questionnaire that reassess cultural humility, cultural awareness and the usability and acceptability of the SE.

Sample: The target population for this study includes undergraduate and graduate nursing students and clinical faculty at Queen's University. A convenience sample of a minimum of 100 nursing students and 20 clinical faculty/clinical instructors will be recruited to participate in this study. Clinical faculty/instructors will be introduced to the study and invited to participate in person during their yearly faculty orientation. Nursing students will be invited to participate via email and in person during their classes.

Setting: The setting will include a University, School of Nursing, in Southern, Ontario, Canada.

Quantitative data will be collected using a web-based survey through Qualtrics©. All participants will assign themselves an ID number (see Appendix for how the ID number will be created).

Participants will be asked to enter this ID number at the beginning of the pre-simulation and post- simulation questionnaires. After providing consent to participate in the study, participants will immediately complete the demographic information and the pre-simulation questionnaire. Once this information has been obtained, they will complete the education session and they will receive an electronic link to the simulation experience (SE) and the post-simulation questionnaire.

Outcome measures: To evaluate usability, engagement, and impact as perceived by participants the ClassRoom Instructional Support Perceptions (CRISP-VS) will be used. The CRISP-VS is 23 item, valid and reliable outcome measure previously used in studies with nursing students.

Reliability testing for the CRISP-VS reports a Cronbach's α of 0.79 for the usability subscale, 0.89 for the engagement subscale, and 0.82 for the impact subscale.

To evaluate cultural humility the Foronda's Cultural Humility Scale will be used. This outcome measure includes 19 questions and was validated and tested with 322 undergraduate nursing and health sciences students and yielded a Cronbach's α = 0.85.

The Foronda Cultural Humility Scale has three subscales including 1) context for difference in perspective; 2) self-attributes; and 3) outcomes of cultural humility. To evaluate cultural awareness the Cultural Diversity Awareness Questionnaire will be used. This questionnaire is designed to measure beliefs and behaviours regarding cultural diversity and inclusion. It is scored by summing the numbers chosen on the questionnaire (1 = never, 2 = almost, 3 = sometimes, 4 = almost always, 5 = always). A high score indicates the individual/participant has a good awareness of their biases and how their behaviours may impact others, the individual relates to others in ways that value diversity. The validity and reliability for the Cultural Diversity Awareness Questionnaire was tested with public school educators and it has a Cronbach's α = 0.9.

Data Analysis: Data will be analyzed using SPSS (IBM, V 29.0.1.1, 2021). Demographic data and the CRISP-VS will be analyzed using descriptive statistics including means, standard deviations and frequencies. To examine if there is a significant difference between pre-simulation and post-simulation cultural humility and cultural awareness scores, paired t-tests will be completed if the data is normally distributed. If the data is not normally distributed a Wilcoxon nonparametric test will be completed. A p- value of 0.05 or less will be considered significant. Reliability testing will also be conducted on the Cultural Diversity Awareness Questionnaire by calculating the Cronbach's α as this outcome measure has not been utilized with the Canadian nursing and nursing student population.

ELIGIBILITY:
Inclusion Criteria:

* undergraduate and graduate nursing students at a University in Southern Ontario
* clinical faculty at a University in Southern Ontario
* speak, read and understand English.
* able to navigate a virtual simulation experience using an electronic device.

Exclusion Criteria:

* students not enrolled in the nursing program
* faculty not teaching in the nursing program

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Cultural Humility | Day 1
  To evaluate cultural humility the Foronda's Cultural Humility Scale will be used. This outcome measure includes 19 questions and was validated and tested with 322 undergraduate nursing and health sciences students and yielded a Cronbach's α = 0.85 (Foronda, Porter & Phitwong, 2021).
  The Foronda Cultural Humility Scale has three subscales including 1) context for difference in perspective; 2) self-attributes; and 3) outcomes of cultural humility.

SECONDARY OUTCOMES:
Cultural Awareness | Day 1
  . To evaluate cultural awareness the Cultural Diversity Awareness Questionnaire will be used (Bennett, 1986, Van Hook, 2000). This questionnaire is designed to measure beliefs and behaviours regarding cultural diversity and inclusion. It is scored by summing the numbers chosen on the questionnaire (1 = never, 2 = almost, 3 = sometimes, 4 = almost always, 5 = always). A high score indicates the individual/participant has a good awareness of their biases and how their behaviours may impact others, the individual relates to others in ways that value diversity (Illinois Leadership Project, 2016). The validity and reliability for the Cultural Diversity Awareness Questionnaire was tested with public school educators and it has a Cronbach's α = 0.9 (Henry, 1995).
usability, engagement, and impact | Day 1
  To evaluate usability, engagement, and impact as perceived by participants the ClassRoom Instructional Support Perceptions (CRISP-VS) will be used. (see Appendix) The CRISP-VS is 23 item, valid and reliable outcome measure previously used in studies with nursing students.
  Reliability testing for the CRISP-VS reports a Cronbach's α of 0.79 for the usability subscale, 0.89 for the engagement subscale, and 0.82 for the impact subscale (Sheng, et al., 2019).

CONTACTS AND LOCATIONS:
Locations (1):
- Queen's University, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li JS, Patterson M, Gumapac NP, Sau C, Mohamed S, Yusef HA, Sawhney M. Simulation Experiences Focusing on Addressing Culturally Based Hidden Bias and RacisM (A-CHARM). J Nurs Educ. 2025 Jul;64(7):449-453. doi: 10.3928/01484834-20240612-04. Epub 2024 Sep 20. PMID 39292736